CLINICAL TRIAL: NCT05956977
Title: Evaluation of 3D Ultrasound in Brain Tumor Surgery
Acronym: Neuro3DUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Collaborators: Brainlab AG (Industry)
Responsible Party: Principal Investigator, Jan Coburger, apl. Prof. Dr. med. Jan Coburger, Consultant, University of Ulm
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuro3DUS
Record Dates: First submitted 2023-04-24; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Residual Tumor
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: retrospective matched pair control
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prospective arm (Experimental): Use of 3D ultrasound intraoperative before intraoperative MRI
  Interventions: Device: resection with help of 3D ultrasound
- retrospective matched pair arm (No Intervention): no use of intraoperative ultrasound before intraoperative MRI

INTERVENTIONS:
Device: resection with help of 3D ultrasound — see above
  Arms: prospective arm

SUMMARY:
Evaluation of impact of use of 3D ultrasound in brain tumor surgery on extend of resection. Benefit for surgery, neurological outcome, accuracy and image quality are secondary outcome parameters. Control group is a retrospective matched pair cohort.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 suspected intra-axial lesion (metastasis or Glioma) potential gross total resection of lesion

Exclusion Criteria:

* no ability for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Extent of resection | 48 hours after surgery
  Volumetric assessment of residual T1 contrast enhancement or FLAIR signal changes in enhancing and non-enhancing glioma, respectively.

SECONDARY OUTCOMES:
image quality | during surgery
  ultrasound image quality, both for 2D and 3D as rated by surgeon and scored from 1(best) to 6 (worst).
neurological outcome | both after surgery and at 3 months
  both at discharge and at 3 months follow up using NIHSS Score
Accuracy of device | during surgery
  ultrasound image acuracy compared to preoperative MRI, both for 2D and 3D as rated by surgeon and scored from 1(best) to 6 (worst), including rating of brainshift and navigation inaccuracy.

OTHER OUTCOMES:
brainshift during surgery | during surgery
  brainshift in mm during surgery comparing preoperative landmarks with intraoperative landmarks in ultrasound and intraooperative MRI

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University of Tübingen, Tübingen, Baden Würtemberg
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aleo D, Elshaer Z, Pfnur A, Schuler PJ, Fontanella MM, Wirtz CR, Pala A, Coburger J. Evaluation of a Navigated 3D Ultrasound Integration for Brain Tumor Surgery: First Results of an Ongoing Prospective Study. Curr Oncol. 2022 Sep 15;29(9):6594-6609. doi: 10.3390/curroncol29090518. PMID 36135087